CLINICAL TRIAL: NCT05823298
Title: Cultural Adaptation of Fugl-Meyer Assessment to Turkish and Evaluation of Psychometric Properties in Acute Stroke Patients
Brief Title: Turkish Adaptation and Psychometric Properties of Fugl-Meyer Assessment in Acute Stroke Patients
Acronym: FMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Zeynep Lide Uz, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: FMA Acute Stroke
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute; Cerebrovascular; Disorder, Acute
Keywords: acute stroke; fugl-meyer assessment; upper extremity; lower extremity; outcome assessment; stroke rehabilitation; translation and cross-cultural adaptation; validity; reliability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this methodological study is to adapt the Fugl-Meyer assessment to Turkish culture and to test its validity and reliability in acute phase stroke patients.

DETAILED DESCRIPTION:
According to the definition of the World Health Organization, stroke is a clinical syndrome that causes rapid focal (or global) cerebral function loss for no apparent reason other than vascular causes, and symptoms persist for more than 24 hours or lead to death.

To effectively manage the post-stroke processes and establish an effective treatment plan, a comprehensive assessment is necessary. One of the most common motor problems following a stroke is hemiplegia, which makes it challenging for the patient to perform activities of daily living and ambulation. Understanding the mechanisms of motor control and motor learning, which are vital components of stroke rehabilitation, necessitates the assessment of motor function. For evaluating motor function in stroke patients, there are numerous outcome measures available. The Fugl-Meyer Assessment (FMA) stands out when comparison of these assessments in terms of clinical and psychometric values. There is no official FMA version that has been translated into Turkish, even though Fugl-Meyer assessment is used in numerous research in Turkey. The aim of this study is to adapt the Fugl-Meyer assessment to Turkish culture and to test its validity and reliability in acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed with stroke
* Less than 1 month passed after onset of stroke
* Upper and lower extremity motor involvement between Brunnstrom stages 2 and 5
* Voluntarily accepting to participate in this research

Exclusion Criteria:

* Visual and hearing impairment
* Upper or lower extremity amputation
* Significant cognitive impairment (Mini Mental State Test Score < 18)
* Mental disorders affecting daily life functioning
* Global aphasia
* Other unstable conditions that may affect participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients who were hospitalized in Istinye University Liv Hospital Brain Angiography Stroke Center between May 2023 to December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | 5 minutes
  a scale used to assess functional independence. Points ranging from 0 to 100.
Modified Rankin Scale | 5 minutes
  a 6 point disability scale with possible scores ranging from 0 to 5

SECONDARY OUTCOMES:
Berg Balance Scale | 10 minutes
  a scale to measure balance in older adults with scores ranging from 0 to 56

CONTACTS AND LOCATIONS:
Overall Officials: Lide Z Uz, 1, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İstinye University Brain Angiography Stroke Center, Istanbul, Esenyurt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baker K, Cano SJ, Playford ED. Outcome measurement in stroke: a scale selection strategy. Stroke. 2011 Jun;42(6):1787-94. doi: 10.1161/STROKEAHA.110.608505. Epub 2011 May 12. PMID 21566236
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Bushnell C, Bettger JP, Cockroft KM, Cramer SC, Edelen MO, Hanley D, Katzan IL, Mattke S, Nilsen DM, Piquado T, Skidmore ER, Wing K, Yenokyan G. Chronic Stroke Outcome Measures for Motor Function Intervention Trials: Expert Panel Recommendations. Circ Cardiovasc Qual Outcomes. 2015 Oct;8(6 Suppl 3):S163-9. doi: 10.1161/CIRCOUTCOMES.115.002098. PMID 26515205
- [Background] Carr JH, Shepherd RB, Nordholm L, Lynne D. Investigation of a new motor assessment scale for stroke patients. Phys Ther. 1985 Feb;65(2):175-80. doi: 10.1093/ptj/65.2.175. PMID 3969398
- [Background] de Vet HC, Terwee CB, Knol DL, Bouter LM. When to use agreement versus reliability measures. J Clin Epidemiol. 2006 Oct;59(10):1033-9. doi: 10.1016/j.jclinepi.2005.10.015. Epub 2006 Aug 10. PMID 16980142
- [Background] Deyo RA, Centor RM. Assessing the responsiveness of functional scales to clinical change: an analogy to diagnostic test performance. J Chronic Dis. 1986;39(11):897-906. doi: 10.1016/0021-9681(86)90038-x. PMID 2947907
- [Background] Duncan PW, Propst M, Nelson SG. Reliability of the Fugl-Meyer assessment of sensorimotor recovery following cerebrovascular accident. Phys Ther. 1983 Oct;63(10):1606-10. doi: 10.1093/ptj/63.10.1606. PMID 6622535
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Gladstone DJ, Danells CJ, Black SE. The fugl-meyer assessment of motor recovery after stroke: a critical review of its measurement properties. Neurorehabil Neural Repair. 2002 Sep;16(3):232-40. doi: 10.1177/154596802401105171. PMID 12234086
- [Background] Malouin F, Pichard L, Bonneau C, Durand A, Corriveau D. Evaluating motor recovery early after stroke: comparison of the Fugl-Meyer Assessment and the Motor Assessment Scale. Arch Phys Med Rehabil. 1994 Nov;75(11):1206-12. doi: 10.1016/0003-9993(94)90006-x. PMID 7979930
- [Background] Mayo NE, Wood-Dauphinee S, Ahmed S, Gordon C, Higgins J, McEwen S, Salbach N. Disablement following stroke. Disabil Rehabil. 1999 May-Jun;21(5-6):258-68. doi: 10.1080/096382899297684. PMID 10381238
- [Background] Alt Murphy M, Resteghini C, Feys P, Lamers I. An overview of systematic reviews on upper extremity outcome measures after stroke. BMC Neurol. 2015 Mar 11;15:29. doi: 10.1186/s12883-015-0292-6. PMID 25880033
- [Background] Salter K, Jutai JW, Teasell R, Foley NC, Bitensky J. Issues for selection of outcome measures in stroke rehabilitation: ICF Body Functions. Disabil Rehabil. 2005 Feb 18;27(4):191-207. doi: 10.1080/09638280400008537. PMID 15824050
- [Background] See J, Dodakian L, Chou C, Chan V, McKenzie A, Reinkensmeyer DJ, Cramer SC. A standardized approach to the Fugl-Meyer assessment and its implications for clinical trials. Neurorehabil Neural Repair. 2013 Oct;27(8):732-41. doi: 10.1177/1545968313491000. Epub 2013 Jun 17. PMID 23774125
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] The World Health Organization MONICA Project (monitoring trends and determinants in cardiovascular disease): a major international collaboration. WHO MONICA Project Principal Investigators. J Clin Epidemiol. 1988;41(2):105-14. doi: 10.1016/0895-4356(88)90084-4. PMID 3335877
- See also: Official Fugl-Meyer Assessment Website — https://www.gu.se/en/neuroscience-physiology/fugl-meyer-assessment